CLINICAL TRIAL: NCT03566953
Title: Dietary Influences On Caries Index Among Sudanese And Egyptian Adult Population A-Cross_Sectional Study
Brief Title: Dietary Influences On Caries Index Among Sudanese And Egyptian Adult Population
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maza Alser Mohamedali, Dietary Influences On Caries Index Among Sudanese And Egyptian Adult Population, Cairo University
Other Study IDs: DIOCIASAEAP-2018
Record Dates: First submitted 2018-06-13; First posted 2018-06-25 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Dental Caries
Keywords: Dental Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the objective of this study is to compare the caries index between Sudanese and Egyptian adult Population in patients with different diet habits and different oral hygiene state in range of (18-40) years old

DETAILED DESCRIPTION:
A main factor for planning any preventive program is to accurately assess a person's risk of developing a caries.

There is a relative lack of data pertaining to adults in the developing world in general and in Sudan in particular. Most of the studies focused on school children.

Many people in Sudan do not receive regular dental care and have acute problems when seen by a dentist. In Sudan the dentist-to-patient ratio is 1:33,000 compared with approximately 1:2,000 in most industrialized countries. Relative to the size of the Sudanese population, there are very few dentists and this restricts access to regular dental care. Other factors which influence dental. Attendance in Sudan include the lack of public funding for oral healthcare and dental insurance schemes to ameliorate the cost of care. For this reason, insufficient awareness of the culture of selecting suitable foods to preserve the health of the mouth and teeth, as prevention is better than treatment .

The study will help the clinician to compare the incidence of caries between different nationality they have different diet habits ,food traditions , and they have different education and cultural levels as these factors can reflect the health care system , and to determine the effect of these factors clearly on dental caries It also allow the clinician to develop the most suitable preventive treatment plan for each patient by evaluating the main causative factor to patient and to eliminate that factor so that we can arrest an ongoing active lesion and prevent developing a new lesion at lowest therapeutic cost.

The patient will be informed in the same visit about the causative factor of the carious lesion in general, the role of diet in particular and instructed about the suggested treatment plan ,to change the lifestyle to the better and strengthen the concept of "prevention is better than treatment"

ELIGIBILITY:
Inclusion Criteria:

* Patients should be in range of 18-40 years old.
* Patient should have good periodontal health.
* Sudanese and Egyptian population

Exclusion Criteria:

* Patient below 18 years and above 40 years old
* Nationality other than Egyptian and Sudanese

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: patient attending Conservative Dentistry department, faculty of dentistry, Cairo University Egypt, will be screened for diagnosis of their chief complaint. Patients will be enrolled in this study if they are compatible with eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dental caries | 3 month
  Caries index(DMFT)

SECONDARY OUTCOMES:
Diet analysis | 3 month
  CAMBRA

CONTACTS AND LOCATIONS:
Overall Officials: Maza Al MohamedAli, master, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moynihan PJ, Kelly SA. Effect on caries of restricting sugars intake: systematic review to inform WHO guidelines. J Dent Res. 2014 Jan;93(1):8-18. doi: 10.1177/0022034513508954. Epub 2013 Dec 9. PMID 24323509